CLINICAL TRIAL: NCT05494216
Title: Advanced Sperm Selection Techniques and Their Contribution to Blastocyst Euploidy Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GFC-005
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Sperm DNA Fragmentation; Infertility
Keywords: Sperm selection; PICSI; MACS; Sperm DNA fragmentation; PGT-A; Euploidy rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICSI (Active Comparator): Semen processing is done by double layer density gradient method followed by adding Sperm to the dot of hyaluronan on the PICSI dish, within minutes the bound sperm are attached by their acrosome to the surface of the dot. Individual bound sperm selection is done followed y ICSI
  Interventions: Other: PICSI
- MACS (Active Comparator): Semen processing is done by double layer density gradient method. The resulted pellet is labeled with annexin V microbeads followed by separation on MACS Column, the eluted fraction contains non apoptotic sperm suitable for ICSI.
  Interventions: Other: MACS

INTERVENTIONS:
Other: PICSI — Sperm selection using PICSI dish for selecting sperm with lower DNA fragmentation index
  Arms: PICSI
Other: MACS — Sperm selection using MACS for selecting sperm with lower DNA fragmentation index
  Arms: MACS

SUMMARY:
Comparing different advanced sperm selection techniques like Physiological ICSI (PICSI) and magnetic activated cell sorting (MACS) in terms of the PGT-A outcomes of each arm blastocysts

DETAILED DESCRIPTION:
Advanced sperm selection methods like PICSI and MACS have been developed for selecting a healthy mature non apoptotic sperm with lower Sperm DNA fragmentation. Previous studies compared the pre-implantation embryo development parameters of those techniques, but none looked at comparing the PGT-A results or euploidy rates of the blastocysts derived from each sperm selection.

PGT-A cases will be randomized on the day of ICSI to the 2 assigned sperm selection techniques.

ELIGIBILITY:
Inclusion Criteria:

* Case must have PGT-A for all of her blastocysts
* Males diagnosed with abnormal sperm DNA fragmentation index (> 20%).
* Normo responder (> 5 mature oocytes)
* Male will have to refrain from ejaculation no less than 1 day but no greater than 3 days prior semen specimen production on day of ICSI

Exclusion Criteria:

* Leukocytospermia
* Presence of varicocele.
* Known genetic abnormality
* Use of sperm or oocyte donors
* Use of gestational carrier
* Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previous uterine infection
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 515 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Euploidy rate | 15 days post ICSI
  Defined as the proportion of euploid blastocysts
Aneuploidy rate | 15 days post ICSI
  Defined as the proportion of aneuploid blastocysts
Low mosaic rate | 15 days post ICSI
  Defined as the proportion of low mosaic blastocysts
High mosaic rate | 15 days post ICSI
  Defined as the proportion of high mosaic blastocysts

SECONDARY OUTCOMES:
Fertilization rate | 1 day
  Defined as the proportion of fertilizaed oocytes
Cleavage rate | 3 days
  Defined as the proportion of cleaved embryos on day 3
Blastocyst development rate | 5-6 days
  Defined as the proportion of blastocysts formed on day 5 or 6
Blastocyst quality rate | 5-6 days
  Defined as the assessment of blastocyst quality according to Gardner's criteria into: good, fair or poor

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hasanen, BSc., Principal Investigator — Ganin Fertility Center; Manar Hozayen, MSc., Principal Investigator — Ganin Fertility Center; Amr Elshimy, BSc., Principal Investigator — Ganin Fertility Center; Hanaa Alkhader, MBBS/MD, Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc, FRCOG, Study Director — Ganin Fertility Center; Yara Hazem, BP, Principal Investigator — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Undecided